CLINICAL TRIAL: NCT03858374
Title: The Design and Application of Air Suspension Biodegradable Patient Transport Pad
Brief Title: Air Suspension Biodegradable Patient Transport Pad
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018PY011
Record Dates: First submitted 2019-02-18; First posted 2019-02-28 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Patients in experimental group were transferred by air-suspending mattress.
  Interventions: Device: transferred by air-suspending mattress
- control group 1 (Active Comparator): Patients in control group 1 were transferred by slide board.
  Interventions: Device: transferred by slide board
- control group 2 (Active Comparator): Patients in control group 2 were transferred by bedsheet.
  Interventions: Device: transferred by bedsheet

INTERVENTIONS:
Device: transferred by air-suspending mattress — Put mattress in advance on the bed. When patients need to be transferred from bed to bed, fill the mattress with gas and keep it inflated, then pull the mattress .
  Arms: Experimental group
Device: transferred by slide board — When patients need to be transferred from bed to bed, insert slide board under patient, then pull the slide board.
  Arms: control group 1
Device: transferred by bedsheet — When patients need to be transferred from bed to bed, just lift the bedsheet.
  Arms: control group 2

SUMMARY:
On the one hand, transferring patient from bed to bed is usually handling by the manual lifting of several staffs or utilizing bedsheet, slide sheet , shovel-style stretcher or other devices to move and lift patients. Whatever, there are some advantages using these devices.

On the other hand, nurses are among the professionals at the highest risk for musculoskeletal disorders. The Bureau of Labor Statistics has shown that overexertion in manual lifting was the main event or exposure leading to injury or illness involving time away from work. Excessive weights, awkward postures, and repetitive motions are some of the known risk factors that contribute to sprains/strains and back injuries. During the process of patient transferring , it refers to the above risk factors for health-care workers. It recommended that using appropriate assistive equipment can reduce the injuries. If staff is safe, patients are safer.

The research team has designed and produced a new transport assistive devices-- biodegradable and air-suspending transfer mattress, which was precisely controlled by gas flow and based on ergonomics. And then apply it to the clinic in order to find whether it's benefit for patients and nursing staff.

It is a randomized controlled trial design.

DETAILED DESCRIPTION:
Research design：randomized controlled trials. Computer generated random numbers. The patients were randomly divided into three groups, ① transfer patients by air-suspending mattress, ② transfer patients by slide board, ③ transfer patients by bedsheets.

Participants: passive patient with transports needs, such as CT/ MRI examination etc. The sample size estimation was according to the formula of multiple parallel design. The main outcome measure was the perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* Passive patient with transfer requirements, such as CT/ MRI examination , transfer from one department to another etc；Patients or their family signed an informed consent.

Exclusion Criteria:

* The patients weighted over 150kg and have spine fracture ；age< 15 years old.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Force value | Day 1
  Spring balance was used to measured the pulling force while transferring patients.(Force value in N)
perceived exertion | Day 1
  Perceived exertion was evaluated by using the Borg Scale of 6-20, which the values near 6 and 20 represent low and high physical exertion, respectively.（perceived exertion in scores）

SECONDARY OUTCOMES:
respiration rate | Day 1（before and after transferring）
  Be recorded by ECG monitor the moment before and after transferring.（respiration rate in bpm）
blood pressure | Day 1（before and after transferring）
  Be recorded by ECG monitor the moment before and after transferring.(blood pressure in mmHg)
heart rate | Day 1（before and after transferring）
  Be recorded by ECG monitor the moment before and after transferring.（heart rate in bpm）
oxygen saturation | Day 1（before and after transferring）
  Be recorded by ECG monitor the moment before and after transferring.
Transfer time | Day 1
  Stopwatch was used to record the time from using the assistive devices to moving the patients to another bed.（transfer time in minutes）

OTHER OUTCOMES:
Satisfaction of patient | Day 1
  Self-made satisfaction questionnaire was used to get the patients' satisfaction about the assistive devices after transferring patients.It includes five items about the feelings of assistive devices while moving--comfort, safety, pain, stability and sound. All the answers take five levels, level five means very satisfied and level one represents very dissatisfied.(Satisfaction of patient in scores)
Satisfaction of nurse staff | Day 1
  Self-made satisfaction questionnaire was used to get nurse staffs' satisfaction about the assistive devices after transferring patients. It includes seven items about using the devices to move patients --no adverse events, saving energy, saving time, convenience, applicability, strong support and total satisfaction. All the answers take five levels, level five means very satisfied and level one represents very dissatisfied.(Satisfaction of patient in scores)

CONTACTS AND LOCATIONS:
Overall Officials: jingfen Jin, Master, Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China